CLINICAL TRIAL: NCT03131219
Title: A Phase 3, Open-Label, Multicenter Study of ALXN1210 in Children and Adolescents With Atypical Hemolytic Uremic Syndrome (aHUS)
Brief Title: Study of Ravulizumab in Children and Adolescents With Atypical Hemolytic Uremic Syndrome (aHUS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1210-aHUS-312; 2016-002499-29 (EudraCT Number)
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Atypical Hemolytic Uremic Syndrome (aHUS)
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome | interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ravulizumab (Experimental): Participants were administered weight-based doses of ravulizumab every 8 weeks thereafter for participants weighing ≥ 20 kg, or once every 4 weeks for participant weighing < 20 kg, for a total of 26 weeks of study treatment in the initial Evaluation Period.
  After the Initial Evaluation Period, participants rolled over into an Extension Period in which all participant continued their weight-based maintenance dose until the product was registered or approved (in accordance with country specific regulation) or for up to 4.5 years, whichever occurred first.
  Interventions: Biological: Ravulizumab

INTERVENTIONS:
Biological: Ravulizumab — Participant received weight-based dosages for 26 weeks during the Initial Evaluation Period. Participants received a loading dose on Day 1, followed by maintenance dosing on Day 15 and once every 8 weeks thereafter for participants weighing ≥ 20 kg, or once every 4 weeks for participant weighing < 20 kg.
  Other Names: ALXN1210; Ultomiris

SUMMARY:
The purpose of the study is to assess the efficacy of ravulizumab to control disease activity in children and adolescents with aHUS who have not previously used a complement inhibitor (complement inhibitor treatment-naïve), as well as in complement inhibitor-experienced (eculizumab-experienced) adolescent participants.

ELIGIBILITY:
Inclusion Criteria:

Complement Inhibitor Treatment Naïve:

1. Participants from birth up to <18 years of age and weighing ≥5 kilograms (kg) at the time of consent.
2. Participants had not been previously treated with complement inhibitors.
3. Evidence of thrombotic microangiopathy (TMA), including low platelet count, hemolysis (breaking of red blood cells inside of blood vessels), and decreased kidney function.
4. Documented meningococcal vaccination not more than 3 years prior to dosing, and vaccination against Streptococcus pneumoniae and Haemophilus influenzae type b.
5. Female participants of childbearing potential and male participants with female partners of childbearing potential must have used highly effective contraception starting at screening and continuing until at least 8 months after the last dose of ravulizumab.

Eculizumab Experienced:

1. Participants between 12 and <18 years of age (non-Japanese sites) or <18 years of age (Japanese sites) who had been treated with eculizumab according to the labelled dosing recommendation for aHUS for at least 90 days prior to screening.
2. Participants with documented diagnosis of aHUS.
3. Participants with clinical evidence of response to eculizumab indicated by stable TMA parameters at screening.
4. Documented meningococcal vaccination not more than 3 years prior to dosing, and vaccination against Streptococcus pneumoniae and Haemophilus influenzae type b.
5. Females of childbearing potential and male participants with female partners of childbearing potential must have used highly effective contraception starting at screening and continuing until at least 8 months after the last dose of ravulizumab.

Exclusion Criteria:

1. Known familial or acquired ADAMTS13 ("a disintegrin and metalloproteinase with a thrombospondin type 1 motif, member 13") deficiency (activity <5%).
2. Known Shiga toxin-related hemolytic uremic syndrome.
3. Positive direct Coombs test.
4. Females who planned to become pregnant during the study or were currently pregnancy or breastfeeding.
5. Identified drug exposure-related hemolytic uremic syndrome.
6. Bone marrow transplant/hematopoietic stem cell transplant within the last 6 months prior to the start of screening.
7. Hemolytic uremic syndrome related to known genetic defects of cobalamin C metabolism.
8. Known systemic sclerosis (scleroderma), systemic lupus erythematosus, or antiphospholipid antibody positivity or syndrome.
9. Chronic dialysis (defined as dialysis on a regular basis as renal replacement therapy for end-stage kidney disease.
10. For eculizumab-experienced participants, prior use of complement inhibitors other than eculizumab.
11. For eculizumab-experienced participants, any known abnormal TMA parameters within 90 days prior to screening.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (6):
  - Research Site, Hollywood, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Detroit, Michigan
  - Research Site, Omaha, Nebraska
  - Research Site, Hackensack, New Jersey
  - Research Site, Charlotte, North Carolina
- Research Site, Brussels, Belgium
- Research Site, Heidelberg, Germany
- Research Site, Milan, Italy
- South Korea (3):
  - Research Site, Jeju-do
  - Research Site, Seoul
  - Research Site, Yangsan
- Spain (4):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Esplugues de Llobregat
  - Research Site, Valencia
- United Kingdom (2):
  - Research Site, Glasgow
  - Research Site, London

REFERENCES:
- [Result] Rondeau E, Scully M, Ariceta G, Barbour T, Cataland S, Heyne N, Miyakawa Y, Ortiz S, Swenson E, Vallee M, Yoon SS, Kavanagh D, Haller H; 311 Study Group. The long-acting C5 inhibitor, Ravulizumab, is effective and safe in adult patients with atypical hemolytic uremic syndrome naive to complement inhibitor treatment. Kidney Int. 2020 Jun;97(6):1287-1296. doi: 10.1016/j.kint.2020.01.035. Epub 2020 Mar 6. PMID 32299680
- [Derived] Dixon BP, Kavanagh D, Aris ADM, Adams B, Kang HG, Wang E, Garlo K, Ogawa M, Amancha P, Chakravarty S, Heyne N, Kim SH, Cataland S, Yoon SS, Miyakawa Y, Luque Y, Muff-Luett M, Tanaka K, Greenbaum LA. Ravulizumab in Atypical Hemolytic Uremic Syndrome: An Analysis of 2-Year Efficacy and Safety Outcomes in 2 Phase 3 Trials. Kidney Med. 2024 Jun 14;6(8):100855. doi: 10.1016/j.xkme.2024.100855. eCollection 2024 Aug. PMID 39105067
- [Derived] Pugh D, O'Sullivan ED, Duthie FA, Masson P, Kavanagh D. Interventions for atypical haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Mar 23;3(3):CD012862. doi: 10.1002/14651858.CD012862.pub2. PMID 33783815
- [Derived] Tanaka K, Adams B, Aris AM, Fujita N, Ogawa M, Ortiz S, Vallee M, Greenbaum LA. The long-acting C5 inhibitor, ravulizumab, is efficacious and safe in pediatric patients with atypical hemolytic uremic syndrome previously treated with eculizumab. Pediatr Nephrol. 2021 Apr;36(4):889-898. doi: 10.1007/s00467-020-04774-2. Epub 2020 Oct 13. PMID 33048203
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1210-aHUS-312&attachmentIdentifier=5ae2d7b1-7696-4a07-bb98-7e5aeac5849c&fileName=ALXN1210-aHUS-312_EOS_Addendum_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Complement Inhibitor Treatment Naïve: Complement inhibitor treatment-naïve participants received weight-based doses of ravulizumab during the 26-week Initial Evaluation Period. After the Initial Evaluation Period, participants rolled over into an Extension Period in which all participants continued their weight-based maintenance dose of ravulizumab.
- Eculizumab Experienced: Eculizumab-experienced participants received weight-based doses of ravulizumab during the 26-week Initial Evaluation Period. After the Initial Evaluation Period, participants rolled over into an Extension Period in which all participants continued their weight-based maintenance dose of ravulizumab.
Period: Initial Evaluation Period
Arm/Group | Complement Inhibitor Treatment Naïve | Eculizumab Experienced
Started | 24 | 10
Received At Least 1 Dose of Study Drug | 24 | 10
Completed | 17 | 10
Not Completed | 7 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Deemed Ineligible Post Treatment | 3 | 0
Not completed — Physician Decision | 1 | 0
Period: Extension Period
Arm/Group | Complement Inhibitor Treatment Naïve | Eculizumab Experienced
Started | 17 | 10
Received At Least 1 Dose of Study Drug | 17 | 10
Completed | 16 | 10
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Complement Inhibitor Treatment Naïve | Eculizumab Experienced | Total
Number analyzed (Participants) | 24 | 10 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.0 (4.79) | 11.0 (4.97) | 8.1 (5.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 1 | 15
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 22 | 9 | 31
  Unknown or Not Reported | 0 | 0 | 0
Baseline Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, and met pre-specified eligibility criteria.
  mL/min/1.73 m^2
    number analyzed (Participants) | 18 | 10 | 28
    (all) | 26.4 (21.17) | 104.90 (29.545) | NA (NA) — This value was not calculated.

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Complement Inhibitor Treatment-naïve Participants With Complete Thrombotic Microangiopathy (TMA) Response at Week 26
Description: Complete TMA response during the 26-week Initial Evaluation Period is a composite outcome measure that required normalization of hematological parameters (platelet count and lactate dehydrogenase [LDH]) and improvement in kidney function (≥25% reduction in serum creatinine from baseline); for participants on dialysis, baseline was established at least 6 days after the end of dialysis. Participants had to meet these criteria for 2 separate assessments obtained at least 4 weeks (28 days) apart, and any measurement in between. To be considered a responder during the 26-week Initial Evaluation Period, the latest time point a participant could first meet the response criteria was 28 days before the Week 26 (Day 183) assessment. Formal statistical comparison analyses were not planned for this study. Percentage based on the responders among treated participants. Confidence interval (CI) based on exact confidence limits using the Clopper Pearson method.
Time Frame: Week 26
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, and met pre-specified eligibility criteria. Here, Overall 'Number of Participants Analyzed' signifies those who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Complement Inhibitor Treatment Naïve
Number analyzed (Participants) | 17
percentage of participants
  Complete TMA response | 77.8 [52.4 to 93.6]
  Platelet count normalization | 94.4 [72.7 to 99.9]
  LDH normalization | 88.9 [65.3 to 98.6]
  ≥ 25% improvement in serum creatinine from baseline | 83.3 [58.6 to 96.4]

2. Secondary Outcome: Time To Complete TMA Response In Complement Inhibitor Treatment-naïve Participants
Description: Participants that did not have a response were censored at the date of last visit or study discontinuation at the time when the analysis was performed. The time to complete TMA Response is reported in days. The time of the event of a confirmed complete TMA response was considered the first time point at which all the criteria for complete TMA response were met. Participants had to meet all complete TMA response criteria at 2 separate assessments obtained at least 4 weeks (28 days) apart, and any measurement in between.
Time Frame: Baseline through at least Week 52 and up to Week 111
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, and met pre-specified eligibility criteria.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Complement Inhibitor Treatment Naïve
Number analyzed (Participants) | 18
days | 30.0 [22.0 to 88.0]

3. Secondary Outcome: Proportion Of Complement Inhibitor Treatment-naïve Participants With Complete TMA Response At Week 52
Description: The proportion of participants considered responders, along with a 2-sided 95% CI based on exact confidence limits using the Clopper Pearson method is reported.
Time Frame: Week 52
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, met pre-specified eligibility criteria, and had evaluable data at specified timepoint. Here, Overall 'Number of Participants Analyzed' signifies those who were evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified categories.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Complement Inhibitor Treatment Naïve
Number analyzed (Participants) | 17
proportion of participants
  Complete TMA responder | 0.882 [0.636 to 0.985]
  Platelet count normalization | 0.882 [0.636 to 0.985]
  LDH normalization | 1.000 [0.805 to 1.000]
  ≥25% improvement in serum creatinine from baseline | 1.000 [0.805 to 1.000]

4. Secondary Outcome: Participants Who Do Not Require Dialysis at Weeks 26 and 52
Description: For participants requiring dialysis within 5 days prior to ALXN1210 treatment initiation, the number of participants no longer requiring dialysis is reported.
Time Frame: Week 26 and Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Complement Inhibitor Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 6 | 0
Participants
  Week 26 | 5 | 0
  Week 52 | 6 | 0

5. Secondary Outcome: Change From Baseline In eGFR At Weeks 26 and 52
Description: Kidney function evaluated by eGFR was summarized at baseline and the Week 26 and Week 52 time points using descriptive statistics for continuous variables for the observed value, as well as the change from baseline. The baseline value was defined as the average of the values from the assessments performed prior to the first study drug infusion (these could include results from Screening and the Day 1 visit). A value of 10 mL/min/1.73 m^2 for eGFR was imputed for participants requiring dialysis for acute kidney injury. The observed value and change from baseline are reported in mL/min/1.73 m^2. An increase indicated improvement in kidney function.
Time Frame: Baseline, Week 26 and Week 52
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, met pre-specified eligibility criteria, and had evaluable data at the specified timepoint (Week 26 or Week 52). Here, Overall 'Number of Participants Analyzed' signifies those who were evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified categories.
Measure: Median (Full Range); unit: mL/min/1.73 m^2
Arm/Group | Complement Inhibitor Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 17 | 10
mL/min/1.73 m^2
  Baseline | 22.0 [10 to 84] | 99.75 [54 to 136.5]
  Change From Baseline at Week 26 | 80.0 [0 to 222] | -2.00 [-94 to 18]
  Change From Baseline at Week 52: number analyzed (Participants) | 16 | 10
  Change From Baseline at Week 52 | 94.0 [10 to 230] | -3.00 [-20 to 9]

6. Secondary Outcome: Participants With Change From Baseline In CKD Stage At Weeks 26 and 52
Description: The CKD stage is presented as the change from baseline in the participants that Improved (excluding those with Stage 1 [normal renal function] at baseline as they cannot improve), Worsened (excluding those with Stage 5 at baseline as they cannot worsen), and Stayed the Same, compared to the CKD stage at baseline. Baseline was derived based on the last available eGFR before starting treatment. Stage 5 was considered the worst category, while Stage 1 was considered the best category. A 2-sided 95% CI for the proportion, based on exact confidence limits using the Clopper-Pearson method, was provided for each category. The CKD stage was classified based on the National Kidney Foundation Chronic Kidney Disease Stage.
Time Frame: Baseline, Week 26, and Week 52
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Complement Inhibitor Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 17 | 10
Participants
  Week 26, Improved | 15 | 0
  Week 26, Worsened | 0 | 3
  Week 26, Stayed the Same | 2 | 7
  Week 52, Improved: number analyzed (Participants) | 16 | 10
  Week 52, Improved | 16 | 0
  Week 52, Worsened: number analyzed (Participants) | 11 | 10
  Week 52, Worsened | 0 | 0
  Week 52, Stayed the Same: number analyzed (Participants) | 16 | 10
  Week 52, Stayed the Same | 0 | 10

7. Secondary Outcome: Change From Baseline In Platelet Count At Weeks 26 and 52
Description: The hematologic TMA parameter of platelet count was summarized at baseline and at Week 26 and Week 52 using descriptive statistics for continuous variables for the change from baseline. Results are reported in platelets*10^9/liter (L) blood.
Time Frame: Baseline, Week 26 and Week 52
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, met pre-specified eligibility criteria, and had evaluable data at the specified time point (Week 26 or Week 52). Here, 'Number Analyzed' signifies participants evaluable for specified categories.
Measure: Median (Full Range); unit: platelets*10^9/L
Arm/Group | Complement Inhibitor Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 18 | 10
platelets*10^9/L
  Baseline | 51.25 [14 to 125] | 281.75 [207 to 415.5]
  Change from Baseline at Week 26 | 247.00 [57.5 to 368.5] | -2.25 [-74.5 to 123.5]
  Change from Baseline at Week 52: number analyzed (Participants) | 17 | 10
  Change from Baseline at Week 52 | 213.00 [19.5 to 471.5] | -34.75 [-109 to 109]

8. Secondary Outcome: Change From Baseline In LDH At Weeks 26 and 52
Description: The hematologic TMA parameter of serum LDH was summarized at baseline and at Week 26 and Week 52 using descriptive statistics for continuous variables for the change from baseline. Results are reported in units (U)/L serum.
Time Frame: Baseline, Week 26 and Week 52
Population: as for outcome 5
Measure: Median (Full Range); unit: U/L
Arm/Group | Complement Inhibitor Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 17 | 10
U/L
  Baseline | 1963.00 [772 to 4985] | 206.50 [138.5 to 356]
  Change From Baseline at Week 26: number analyzed (Participants) | 16 | 10
  Change From Baseline at Week 26 | -1851.50 [-4713 to -513] | -8.50 [-50.5 to 50.5]
  Change From Baseline at Week 52: number analyzed (Participants) | 16 | 10
  Change From Baseline at Week 52 | -1825.50 [-4724 to -579] | -17.50 [-34.5 to 29.5]

9. Secondary Outcome: Change From Baseline In Hemoglobin At Weeks 26 and 52
Description: The hematologic TMA parameter of hemoglobin level was summarized at baseline and at Week 26 and Week 52 using descriptive statistics for continuous variables for the change from baseline. Results are reported in grams (g)/L blood.
Time Frame: Baseline, Week 26 and Week 52
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, met pre-specified eligibility criteria, and had evaluable data at the specified timepoint (Week 26 or Week 52). Here, 'Number Analyzed' signifies participants evaluable for specified categories.
Measure: Median (Full Range); unit: g/L
Arm/Group | Complement Inhibitor Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 18 | 10
g/L
  Baseline | 74.25 [32 to 106] | 132.00 [114.5 to 148]
  Change From Baseline at Week 26: number analyzed (Participants) | 15 | 10
  Change From Baseline at Week 26 | 46.50 [26.5 to 86] | -3.50 [-19.5 to 8]
  Change From Baseline at Week 52: number analyzed (Participants) | 17 | 10
  Change From Baseline at Week 52 | 51.50 [-19 to 80] | 5.50 [-7.5 to 13.5]

10. Secondary Outcome: Percentage Of Complement Inhibitor Treatment-naïve Participants With An Increase From Baseline In Hemoglobin ≥20 g/L Through Week 26 and Week 52
Description: The percentage of participants with an increase from baseline in hemoglobin ≥20 g/L, observed at 2 separate assessments obtained at least 4 weeks (28 days) apart, and any measurement in between, was assessed through Week 26 and Week 52 and is presented as the percentage of responders, along with a 2-sided 95% CI. The 95% CIs are based on exact confidence limits using the Clopper-Pearson method. To be considered a responder during the 26-week and 52-week Extension Periods, the latest time point a participant could first meet the response criteria was 28 days before the respective Week 26 and Week 52 assessments (components of the response maintained for at least 28 days).
Time Frame: Baseline through Week 26 and through Week 52
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, met pre-specified eligibility criteria, and had evaluable data at the specified timepoints (Week 26 or Week 52). Here, Overall 'Number of Participants Analyzed' signifies those who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Complement Inhibitor Treatment Naïve
Number analyzed (Participants) | 17
percentage of participants
  Week 26 | 100 [80.5 to 100]
  Week 52 | 94.1 [71.3 to 99.9]

11. Secondary Outcome: Change From Baseline In Quality Of Life As Measured By The Functional Assessment Of Chronic Illness Therapy (FACIT)-Fatigue Version 4 Questionnaire (Participants ≥5 Years Of Age) At Weeks 26 and 52
Description: Quality of life was assessed in participants >5 years of age by the Pediatric FACIT-Fatigue Questionnaire (reported by participants who were ≥8 years of age at the time of enrollment; caregiver reported or caregiver assistance for participants who were 5 to <8 years of age at the time of enrollment). The FACIT Fatigue data were summarized at baseline and each post baseline time point using descriptive statistics for continuous variables for the observed value as well as the change from baseline. The FACIT Fatigue Version 4 questionnaire at baseline and each post-infusion time point was scored using standard scoring algorithms. The score ranges from 0 to 52, with a higher score indicating less fatigue. An increase in score indicated an improvement in quality of life.
Time Frame: Baseline, Week 26 and Week 52
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, met pre-specified eligibility criteria, and had evaluable data at the specified timepoint (Week 26 or Week 52). Here, Overall 'Number of Participants Analyzed' signifies those who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Complement Inhibitor Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 9 | 8
units on a scale
  Baseline | 35.00 [4 to 44] | 50.00 [42 to 52]
  Change From Baseline at Week 26 | 10.00 [4 to 48] | 0.00 [-5 to 3]
  Change From Baseline at Week 52 | 9.00 [3 to 47] | -1.00 [-7 to 2]

ADVERSE EVENTS:
Time Frame: From the beginning of the initial evaluation period (Day 1) through data cutoff (at least 52 weeks and up to a maximum of 111 weeks of treatment, representing 36.2 patient-years of exposure).
Arm/Group | Complement Inhibitor Treatment Naïve | Eculizumab Experienced
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/10
Serious Adverse Events (participants affected / at risk) | 16/24 | 1/10
Other Adverse Events (participants affected / at risk) | 21/24 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Complement Inhibitor Treatment Naïve (N=24) | Eculizumab Experienced (N=10)
Gastroenteritis viral (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 1
Cytomegalovirus enteritis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia pyelonephritis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0
Human bocavirus infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Hypertensive urgency (Vascular disorders) | 1 | 0
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Complement Inhibitor Treatment Naïve (N=24) | Eculizumab Experienced (N=10)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 4 (16)
Nasopharyngitis (Infections and infestations) | 7 (13) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (4) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (4)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (9) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (9) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (24) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 1 (1)
Influenza A virus test positive (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 7 (18) | 1 (1)
Asteatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 6 (7) | 1 (1)
Tonsilitis (Infections and infestations) | 3 (4) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (9) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 10 (21) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (8) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vitamin D decreased (Investigations) | 3 (5) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Device occlusion (Product Issues) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT03131219/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT03131219/SAP_001.pdf